CLINICAL TRIAL: NCT00921713
Title: Testing an Optimal Model of Patient-Centered Cancer Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1P20CA137219NN; 1P20CA137219 (NIH)
Record Dates: First submitted 2009-06-04; First posted 2009-06-16 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Cancer
Keywords: Early cancer care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Usual Care (Active Comparator): An extensive packet of information including cancer education materials and treatment resources will be mailed to patients.
  Interventions: Other: Patient-centered materials
- Oncology Nurse Care Management (Experimental): In addition to this mailed information packet, patients in OCNM will be contacted by an experienced Oncology nurse with additional training in self-management support and psychosocial care. The intervention nurse, supported by a Medical Oncologist and Clinical Psychologist, will work closely with patients, their primary care physicians, and other clinicians to assure that patient needs discussed are met. The nurses will be trained in and employ proven counseling and psychotherapeutic approaches-behavioral activation and problem-solving treatment. The multi-component intervention will be based on the Chronic Care Model's six elements (health care organization, community resources, self-management support, delivery system design, decision support, and clinical information system).
  Interventions: Other: Oncology Nurse Care Management

INTERVENTIONS:
Other: Oncology Nurse Care Management
  Arms: Oncology Nurse Care Management
Other: Patient-centered materials
  Arms: Enhanced Usual Care

SUMMARY:
The purpose of this proposal is to develop and test the efficacy in a randomized, controlled clinical trial of an Oncology Nurse Care Management (ONCM) program to support cancer patients early in their course. The ONCM program will be compared with an Enhanced Usual Care (EUC) program that will provide education materials and treatment resources for patients. Efficacy will be measured by differences over time in participant-reported Quality of Life, Symptoms and Emotional Distress, and Quality of Care between patients receiving ONCM versus EUC.

DETAILED DESCRIPTION:
Overall Goal:

Our primary goal is to assess the impact on quality of life, quality of care, and other outcomes of two programs designed to support patients newly diagnosed with breast, colorectal, and lung cancer patients. The Oncology Nurse Care Management (ONCM) and Enhanced Usual Care (EUC) interventions will be implemented and evaluated among enrollees of Group Health.

Specific Aims:

A.1. To develop a robust early cancer notification system based on automated data to facilitate intervention shortly after cancer diagnosis.

A.2. To implement an Oncology Nurse Care Management program that addresses patient questions, symptoms, psychosocial needs, and facilitates timely, coordinated care.

A.3. To compare the impact of the Oncology Nurse Care Manager Program with Enhanced Usual Care in Group Health cancer patients using a randomized clinical trial design. Our two primary outcomes are quality of life and patients' perspectives of quality of care. As secondary outcomes, we will evaluate the impact of the intervention on psychosocial distress and depression.

ELIGIBILITY:
Inclusion Criteria:

1. On the panel of an eligible and consenting primary care physician;
2. Diagnosed with a new occurrence of breast (females only) , colorectal, or lung cancer within the past three weeks;
3. Age 18 or older; and
4. Able to complete the baseline questionnaire.

Exclusion Criteria:

1. They plan to disenroll from GH or be out of the area in the coming year; or
2. Primary care physician or specialty physician expects survival to be less than 12 months; or
3. Don't speak English; or
4. Have moderate cognitive impairment (a score of 3 or more on a six-item validated instrument, or psychosis as assessed by ICD-9 codes from GH medical record data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-09; Primary Completion 2011-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Quality of life and satisfaction with care between patients in Oncology Nurse Care Management versus Enhanced Usual Care | 5/2009 - 8/2011

SECONDARY OUTCOMES:
Treatment adherence and treatment outcomes of patients in Oncology Nurse Care Management versus Enhanced Usual Care | 5/2009 - 8/2011

CONTACTS AND LOCATIONS:
Overall Officials: Edward Wagner, MD, MPH, Principal Investigator — Group Health Research Institute